CLINICAL TRIAL: NCT05800756
Title: Pyrotinib Combined With Trastuzumab, Dalpiciclibe and Letrozole for HR+/HER2+ Breast Cancer:A Single Arm, Open Label, Phase II Trial
Brief Title: Pyrotinib Combined With Trastuzumab,Dalpiciclib and Letrozole for HR+/HER2+ Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-080
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; CDK4/6 inhibitor; hormone receptor-positive; HER2 positive; dalpiciclib; pyrotinib ;
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort 1 (Experimental): patients with stage II-III HR+/HER2+ breast cancer
  Interventions: Drug: pyrotinib combined with trastuzumab, dalpiciclib and letrozole

INTERVENTIONS:
Drug: pyrotinib combined with trastuzumab, dalpiciclib and letrozole — Six 4-week cycles of dalpiciclib orally, 125mg, day 1-21, and letrozole orally, 2.5 mg, day 1-28, and pyrotinib orally, 320mg, day 1-28, and trastuzumab, injection, 8 mg/kg loading dose in cycle 1, 6mg/kg in cycles 2-6, intravenous drops, 1 cycle on day 1-21.

SUMMARY:
In this single arm, open label, phase 2 trial, operable patients with stage II-III HR+/HER2+ breast cancer will be enrolled and receive two cycles of pyrotinib combined with trastuzumab, dalpiciclib and letrozole. Imaging evaluation was performed two weeks later, and patients who achieved CR or PR were continued with the original regimen for 4 cycles. Subjects who did not achieve PR switched to regimen and received 4 cycles of pyrotinib combined with trastuzumab plus chemotherapy. This study aims to assessed the biological effects and safety of pyrotinib combined with trastuzumab, dalpiciclib and letrozole for HR+/HER2+ breast cancer in the neoadjuvant setting.

DETAILED DESCRIPTION:
This is a single arm, open label, phase 2 trial aimed to investigate the biological effects and safety of pyrotinib combined with trastuzumab, dalpiciclib and letrozole for HR+/HER2+ breast cancer. A total of 30 patients with stage II-III HR+/HER2+ breast cancer will be enrolled. Subjects will be enrolled and receive two cycles of pyrotinib combined with trastuzumab, dalpiciclib and letrozole. Imaging evaluation was performed two weeks later, and patients who achieved CR or PR were continued with the original regimen for 4 cycles. Subjects who did not achieve PR switched to regimen and received 4 cycles of pyrotinib combined with trastuzumab plus chemotherapy. In a specific medication cycle, patients use dalpiciclib orally, 125mg, day 1-21, and letrozole orally, 2.5 mg, day 1-28, and pyrotinib orally, 320mg, day 1-28, and trastuzumab, injection, 8 mg/kg loading dose in cycle 1, 6mg/kg in cycles 2-6, intravenous drops, 1 cycle on day 1-21. Premenopausal or perimenopausal patients should combine ovarian function suppression, including bilateral oophorectomy or treatment with gonadotropin-releasing hormone agonists. The primary endpoint is pathological complete response rate. The secondary endpoints include overall response rate, breast-conserving surgery rate and safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. A ECOG PS score of 0-1;
2. Postmenopausal or pre menopausal/perimenopausal women aged ≥ 18 years who must receive LHRH agonists during the study period;
3. Pathological examination confirmed invasive breast cancer with positive ER, PR and HER 2;

(1)Follow the 2018 ASCO-CAP HER 2 positive interpretation guidelines. The pathology laboratory confirms that the immunohistochemical (IHC) score is 3+, or 2+and the in situ hybridization (ISH) test is positive; (2)ER positive was defined as the percentage of ER positive cells ≥ 10%; (3)The percentage of PR positive cells ≥ 10%; 4、The tumor stage is early (T2-3, N0-1, M0) or locally advanced (T2-3, N2-3, M0) patients with breast cancer newly treated; 5、The functions of main organs meet the following requirements (no blood transfusion, no use of whitening and platelet raising drugs within 2 weeks before screening):

1. Blood routine examination: neutrophil (ANC) ≥ 1.5 × 109/L； Platelet count (PLT) ≥ 90 × 109/L； Hemoglobin (Hb) ≥ 90g/L;
2. Blood biochemistry: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN； Alkaline phosphatase ≤ 2.5 × ULN； Urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN；
3. Color Doppler echocardiography: left ventricular ejection fraction (LVEF) ≥ 55%; (4)12 lead ECG: Fridericia corrected QT interval (QTcF)<470 msec. 6、Women who can accept biopsy; 7、Volunteered to participate in this study; signed informed consent; with good compliance and willingness to follow-up.

Exclusion Criteria:

1. Patients with stage IV breast cancer;
2. Inflammatory breast cancer;
3. Previous antineoplastic treatment or radiotherapy for any malignant tumor, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma;
4. At the same time, he received anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy;
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not completely recovered from such surgical procedures;
6. Serious heart disease or discomfort, including but not limited to the following diseases:

(1)History of diagnosis of heart failure or systolic dysfunction (LVEF<50%); (2)High risk uncontrolled arrhythmia, such as atrial tachycardia, resting heart rate>100 bpm, significant ventricular arrhythmia (such as ventricular tachycardia) or higher grade atrioventricular block (i.e. Mobitz Ⅱ second degree atrioventricular block or third degree atrioventricular block); (3)Angina pectoris requiring anti angina drugs; (4)Valvular heart disease with clinical significance; (5)ECG showed transmural myocardial infarction; (6)Poor control of hypertension (systolic blood pressure>180mmHg and/or diastolic blood pressure>100mmHg); 7、Inability to swallow, intestinal obstruction or other factors affecting drug administration and absorption; 8、People known to have a history of allergy to the drug components of this protocol; 9、Have a history of immunodeficiency, including HIV test positive, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; 10、Female patients during pregnancy and lactation, female patients with fertility and positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period and within 7 months after the last study drug use; 11、Those who have a history of abuse of psychotropic substances and cannot quit or have mental disorders; 12、Suffering from serious concomitant diseases or other conditions that may interfere with the planned treatment of concomitant diseases, or any other conditions that the investigator believes are not suitable for the patient to participate in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | up 2 years
  After neoadjuvant therapy, there are no residual invasive tumors in the primary focus and regional lymph nodes of breast cancer, but ductal carcinoma in situ may be present(ypT0/is ypN0)

SECONDARY OUTCOMES:
objective response rate | up 2 years
  The rate of CR and PR,determined using RECIST v1.1 criteria
breast-conserving surgery rate | up 2 years
  The number of cases that actually underwent breast-conserving surgery after surgery accounted for the percentage of all breast cancer patients who underwent surgery
safety profile | up 2 years
  Adverse events (AE) and severe adverse events (SAEs) are recorded. Refer to NCI-CTC AE 5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Guangdong Qiao, Principal Investigator — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China